CLINICAL TRIAL: NCT06802679
Title: Comparison of Standard Versus High Dose Urokinase for Dysfunctional Tunneled Dialysis Catheters in Haemodialysis Patients: a Randomized Controlled Trial
Acronym: SHUT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Healthcare Group, Singapore (Other Government)
Responsible Party: Principal Investigator, Allen Liu Yan Lun, Senior Consultant, National Healthcare Group, Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEG2007; Comparison of Standard versus (Other Grant/Funding Number: Alexandra Health Fund)
Record Dates: First submitted 2025-01-26; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Hemodialysis; Thrombolytic Therapy; Dialysis Access Dysfunction; Randomised Controlled Trial; End Stage Renal Disease (ESRD)
Keywords: urokinase
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIgh dose urokinase (Active Comparator): Patients will be assessed for eligibility for study by nephrologist on duty who is also a PI or Co-I.
  Patients who meet inclusion criteria will be enrolled in study and informed consent taken.
  A trained HD nurse will test the catheter of the patient presenting with TDC dysfunction.
  Once TDC dysfunction is confirmed, patients will be randomized to one of 2 groups and urokinase instillation done according to protocol (see section F9) After a minimum dwell time of 2 hours, urokinase is aspirated and catheter tested by a trained HD nurse. Haemodialysis is then carried out via the catheter.
  Baseline clinical data, urokinase and hemodialysis details will be recorded for each patient visit as per data collection template.
  Interventions: Drug: Urokinase
- Standard dose urokinase (Placebo Comparator): same as above but with different dosage of urokinase
  Interventions: Drug: Urokinase

INTERVENTIONS:
Drug: Urokinase — In the higher dose group: 30,000unit (1.5ml) per catheter lumen is instilled per catheter lumen (in both arterial and venous ports respectively). This allows utilization of the entire vial of Urokinase to prevent wastage and to assess if this increase in dose improves catheter patency and survival, thus reducing the need for a TDC exchange in our HD patients. The urokinase lock is dwelled for at least 2 hours, after which aspiration and catheter testing will be done by a trained HD nurse.
  Other Names: High dose urokinase
  Arms: HIgh dose urokinase
Drug: Urokinase — 20,000unit (1ml) is instilled per catheter lumen (in both arterial and venous ports respectively); and the remaining 1ml is discarded.
  Other Names: Standard dose urokinase
  Arms: Standard dose urokinase

SUMMARY:
Tunneled dialysis catheters (TDCs) remain a frequent form of vascular access for patients undergoing long-term haemodialysis (HD). In our local setting, thrombolytic therapy with urokinase is used as first line therapy to restore catheter patency in patients who develop TDC dysfunction before considering a TDC exchange which is more invasive, requires hospital admission, and involves a higher cost. There are no published local data on the efficacy of Urokinase, though this is widely used in local practice as first line in the management of TDC dysfunction. Previous studies have also varied in terms of study methodology, dose and administration of urokinase in the form of systemic infusion or catheter lock therapy, with varying success rates of 78-97% (2,4-8). Overall, majority of these studies utilized higher doses of urokinase - some studies reported higher patency rates with high dose systemic infusion (4,5) or higher success rates when a higher dose was compared to a lower dose of urokinase lock (6-8). Bleeding events were very rare even in studies that use much higher doses or systemic infusion of urokinase (2,4-8). Our own preliminary data show lower lower success rates of around 52.5% compared to published reports, the question remains on how we can improve our patency rate and cost-effectiveness in treating TDC dysfunction without an increase in risk of adverse events. Therefore, we aim to answer the question as to whether an increase in dose of urokinase will achieve the above outcomes and result in a reduced need for TDC exchange.

ELIGIBILITY:
Inclusion Criteria:

All HD patients aged 21 or above with TDC dysfunction and able to provide informed consent and do not meet any exclusion criteria are eligible for enrolment in the study.

Catheters eligible for the study include:

(i) Incident catheters that have never received urokinase; including newly inserted catheters for previously enrolled patients are allowed.

(ii) Prevalent catheters that have not received urokinase for the last 6 months

Exclusion Criteria:

* Patients with TDC non-function, defined as no inflow and outflow from both arterial and venous ports upon catheter testing.
* Patients with contraindications to Urokinase including active internal bleeding; recent cerebrovascular accident (< 2 months); recent intracranial or intraspinal surgery (< 2 months); intracranial neoplasm, aneurysm or arteriovenous malformation; recent trauma, including cardiopulmonary resuscitation; recent gastrointestinal bleeding (<2 months); known bleeding diathesis; severe uncontrolled hypertension; known hypersensitivity to Urokinase or any ingredient present in its formulation.
* Pregnancy.
* Tunneled dialysis catheter-related blood stream infection

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-01-04 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Primary catheter patency, TDC exchange rate for all visits | 6 months
  Catheter patency right after urokinase aspiration as tested by trained HD nurse (complete / partial / failed) for each patient visit.
  Primary patency: Interval between primary intervention (high versus standard dose urokinase) and repeated intervention for recurring dysfunction in a catheter

SECONDARY OUTCOMES:
Secondary catheter patency, adverse events | 6 months
  Secondary patency: Interval between second episode of dysfunction until TDC exchange / removal or other censorship event achieved (death, change of modality)

CONTACTS AND LOCATIONS:
Locations (1):
- Khoo Teck Puat Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang DH, Mammadov K, Hickethier T, Borggrefe J, Hellmich M, Maintz D, Kabbasch C. Fibrin sheaths in central venous port catheters: treatment with low-dose, single injection of urokinase on an outpatient basis. Ther Clin Risk Manag. 2017 Jan 24;13:111-115. doi: 10.2147/TCRM.S125130. eCollection 2017. PMID 28182117
- [Background] Li Cavoli G, Schillaci O, Zagarrigo C, Servillo F, Li Cavoli TV, Palmeri M, Rotolo U. The urokinase lock-therapy for hemodialysis occluded central venous catheters. Blood Purif. 2015;39(1-3):238. doi: 10.1159/000381007. No abstract available. PMID 25823425
- [Background] Donati G, Coli L, Cianciolo G, La Manna G, Cuna V, Montanari M, Gozzetti F, Stefoni S. Thrombosis of tunneled-cuffed hemodialysis catheters: treatment with high-dose urokinase lock therapy. Artif Organs. 2012 Jan;36(1):21-8. doi: 10.1111/j.1525-1594.2011.01290.x. Epub 2011 Aug 16. PMID 21848863
- [Background] Shavit L, Lifschitz M, Plaksin J, Grenader T, Slotki I. High dose urokinase for restoration of patency of occluded permanent central venous catheters in hemodialysis patients. Clin Nephrol. 2010 Oct;74(4):297-302. doi: 10.5414/cnp74297. PMID 20875382
- [Background] Twardowski ZJ. High-dose intradialytic urokinase to restore the patency of permanent central vein hemodialysis catheters. Am J Kidney Dis. 1998 May;31(5):841-7. doi: 10.1016/s0272-6386(98)70054-x. PMID 9590195
- [Background] Clase CM, Crowther MA, Ingram AJ, Cina CS. Thrombolysis for restoration of patency to haemodialysis central venous catheters: a systematic review. J Thromb Thrombolysis. 2001 Apr;11(2):127-36. doi: 10.1023/a:1011272632286. PMID 11406727
- [Background] Mokrzycki MH, Lok CE. Traditional and non-traditional strategies to optimize catheter function: go with more flow. Kidney Int. 2010 Dec;78(12):1218-31. doi: 10.1038/ki.2010.332. Epub 2010 Sep 29. PMID 20881943
- [Background] Mendes ML, Barretti P, da Silva TN, Ponce D. Approach to thrombotic occlusion related to long-term catheters of hemodialysis patients: a narrative review. J Bras Nefrol. 2015 Apr-Jun;37(2):221-7. doi: 10.5935/0101-2800.20150035. English, Portuguese. PMID 26154643